CLINICAL TRIAL: NCT02594579
Title: Effect of High Dose Vitamin D3 Supplementation on Skeletal Muscle Mass and Body Compositions in Critically Ill Patients With Vitamin D Deficiency
Brief Title: Effect of Vitamin D3 Supplementation on Muscle Mass in ICU Patient
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 075802
Record Dates: First submitted 2015-10-05; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Vitamin D Deficiency; Sarcopenia; Critical Illness
MeSH Terms: conditions — Vitamin D Deficiency; Sarcopenia; Critical Illness | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator): Dietary Supplement: Vitamin D3
  Interventions: Drug: Vitamin D3
- Placebo (Placebo Comparator): Dietary Supplement: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3 100,000 u per day on day 1,3 then 50,000 u/day on day 5,7,9,12 and continue 50,000 u 3 times/ week for 4 weeks
  Other Names: Cholecalciferol (D3-50)
  Arms: Vitamin D
Drug: Placebo — Placebo on day 1,3,5,7,9,12 then 3 times/ week for 4 weeks
  Other Names: Cholecalciferol (D3-50) placebo
  Arms: Placebo

SUMMARY:
A randomized double blind placebo control trial study will be conducted in critically ill patients with vitamin D deficiency. Investigator aimed to study the effect of oral vitamin D3 supplementation, compare to placebo, on skeletal muscle mass and body composition.

DETAILED DESCRIPTION:
There is a high prevalence of vitamin D deficiency in critically ill patient which is associated with muscle wasting and physical disability. Recent study showed that treatment of vitamin D deficiency with high dose vitamin D improved muscle wasting and may prevent further muscle breakdown.

Investigator want to explore whether a high dose vitamin D3 supplementation, compare to placebo will be able to improve muscle wasting in critically ill patients.

The eligible participant will be asked to sign and date the informed consent document then they will be randomized to receive vitamin D3 supplement or placebo, using the computer generated code in conceal envelope.

Vitamin D3 or placebo will be given orally or feeding tube via feeding tube at a dose of 100,000 IU on day 1 and 3 then 50,000 IU on day 5,7,9,12 followed by 150,000 unit per week for 4 week.

Serum 25-Hydroxyvitamin D, 1,25-dihydroxyvitamin D will be measured at baseline (day 0) then day 10 and day 43 after vitamin D supplementation. Moreover, Investigator will assess the diameter of rectus femoris by using ultrasonography on day 0,10 and 43.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70 years old
* Expected ICU stay ≥ 48 hrs

Exclusion Criteria:

* Participate in other clinical trial
* Contraindication to receive oral or enteral feeding
* Do not resuscitate /imminent death
* Vegetative state, generalize weakness, denervation of leg, both leg amputation
* Hypercalcemia or Hypercalcemia at risk
* Hyperphosphatemia,
* History of nephrolithiasis
* End stage renal disease on renal replacement therapy
* Pregnancy/lactation
* Consent refusal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Rectus femoris cross-sectional diameer | Change from baseline Rectus femoris cross-sectional diameter at day 43
  A difference of change from baseline Rectus femoris cross-sectional diameter at day 43 in participant who receive cholecalciferol or placebo

SECONDARY OUTCOMES:
Length of hospital stays | An expected average of 3 weeks
  Participant will be followed for the duration of hospital stay
Length of ICU stays | An expected average of 2 weeks
  Participant will be followed for the duration of ICU stay
Percentage of skeletal muscle mass | Change from basline percentage skeletal muscle mass at day 43
  Percentage of skeletal muscle mass will be assessed using bioelectrical impedance analysis
Correction vitamin D deficiency | 43 days
  Number percentage of participant who above 25(OH)D concentration above or equal 30 in participant who receive cholecalciferol or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Daruneewan Warodomwichit, Principal Investigator — Division of Nutrition and Biochemical medicine, Department of Medicine, Faculty of medicine, Ramathibodi Hospital, Mahidol University Bangkok, Thailand
Locations (1):
- Department of Medicine, Faculty of medicine, Ramathibodi Hospital, Bangkok, Thailand